CLINICAL TRIAL: NCT03940131
Title: Re-challenge Therapy With Chemotherapy and Panitumumab in Metastatic Colorectal Cancer Patients Treated With an Anti-EGFR Therapy in 1st Line Treatment: a Phase II Multicentre Study.
Brief Title: Re-challenge Therapy With Chemotherapy & Panitumumab in Metastatic Colorectal Cancer Patients Treated With an Anti-EGFR
Acronym: REPAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah Medical City (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-504
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: re-challenge; panitumumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Folfox protocol; IFL protocol

STUDY DESIGN:
Intervention Model Description: Single arm Phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Panitumumab with FOLFOX6/FOLFIRI
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — FOLFOX6 regimen consists of 2-hour infusion of oxaliplatin (85 mg/m2) and 2-hour infusion of leucovorin (400 mg/m2 ) on Day l, followed by 5-fluorouracil bolus (400 mg/m2) on Day 1 and 46-hour infusion (2.4 g/m2). FOLFOX6 regimen will be repeated at 2-week intervals. FOLFIRI regimen consists of 2-hour infusion of irinotecan (180 mg/m2) and 2-hour infusion of leucovorin (400 mg/m2 ) on Day l, followed by 5-fluorouracil bolus (400 mg/m2) on Day 1 and 46-hour infusion (2.4 g/m2). FOLFIRI regimen will be repeated at 2-week intervals.
  Other Names: Folfox; Folfiri

SUMMARY:
patients with metastatic colorectal cancer who were initially RAS wild and failed at least 2 lines of chemotherapy will be enrolled. Anti-EGFR must have been given in 1st line. Those who remain RAS-wild upon retesting will receive rechallenge with panitumumab and chemotherapy

DETAILED DESCRIPTION:
This is a single arm pilot multicenter prospective study. We will recruit KRAS/RAS wild metastatic colorectal cancer patients who received at least 2 lines of chemotherapy and the 1st line must include cetuximab/panitumumab combined with chemotherapy. We will repeat RAS testing after progression on the last line of therapy. RAS testing will be taken via liquid biopsy using ctDNA or tissue biopsy from either a new tumour lesion or a previously present lesion which shows evidence of disease progression by radiological imaging. Only RAS-wild patients upon re-testing will be enrolled and will receive re-challenge therapy with panitumumab combined with chemotherapy similar to that given at 1st line (5-fluorouracil/leucoverin combined with oxaliplatin or irinotecan). Those converted to RAS mutant will not be enrolled.

All patients will be treated until disease progression, unacceptable toxic effects or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the colon or rectum with initially KRAS/RAS wild tumours.
* Patients received at least 2 lines of chemotherapy including a fluoropyrimidine, irinotecan and oxaliplatin± bevacizumab.
* First line chemotherapy regimen with a fluoropyrimidine and irinotecan or fluoropyrimidine and oxaliplatin in addition to an anti-EGFR agent (cetuximab/panitumumab).
* No evidence of disease progression for at least 4 months from the start of 1st line therapy.
* At least one measurable lesion ≥ 10 mm as assessed by CT-scan or MRI must be available and accessible for re-biopsy and RAS testing.
* Repeated RAS testing before re-challenge therapy must be done.
* Age ≥18 years.
* ECOG Performance status (PS) 0-2.
* The patient has adequate organ function, defined as : Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, hemoglobin ≥ 9 g/dl, and platelets ≥ 100 x 109/L. Total bilirubin ≤ 1.5 times upper limit of normal value (ULN), serum alkaline phosphatase level < 5 times ULN, Serum creatinine level <1.5 mg/dl.
* For female patients of childbearing potential, negative pregnancy test within 7 days before starting the study treatment.
* Subject must provide informed consent prior to initiation of any study specific activities/procedures

Exclusion Criteria:

* Significant cardiovascular disease including unstable angina or myocardial infarction within 12 months before initiation of study treatment or a history of ventricular arrhythmia (treated or not).
* History or evidence of central nervous system metastasis (CT-scan or MRI are not mandatory if no clinical symptoms).
* Known allergy or hypersensitivity to panitumumab.
* Patients with right-sided colon cancer originating from the ascending colon or hepatic flexure.
* Patients with known MSI-high status.
* Patients with known HER2-positive status.
* Previous or concurrent malignancy except for basal or squamous cell skin cancer, in situ carcinoma of the cervix, low-risk prostate cancer according to d'Amico classification or other solid tumors treated curatively and without evidence of recurrence for at least 5 years prior to the study.
* Active or uncontrolled clinically serious infection.
* Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness.
* Other serious and uncontrolled non-malignant disease.
* Pregnancy.
* Breast feeding.
* Treatment with any other investigational medicinal product within 28 days prior to study entry.
* Concomitant administration of live, attenuated virus vaccine such as yellow fever vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 years
  defined as the proportion of patients with tumour response (complete response or partial response) by RECIST criteria 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 3 years
  defined as the proportion of patients with tumour response (complete response or partial response) or tumour stabilization during study treatment.
Progression-free survival (PFS) | 3 years
  defined as the time from the date of starting the study treatment regimen till the date of the first disease progression after re-challenge therapy or death (any cause).
Overall survival (OS) | 3 years
  defined as the time from the date of starting the study treatment regimen to the date of patient death, due to any cause, or to the last date at which the patient was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Shereef A Elsamany, MD, Principal Investigator — King Abdullah Medical City
Locations (1):
- King Abdullah Medical City, Holy Capital, Mecca, Makkah Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No